CLINICAL TRIAL: NCT02253459
Title: Phase III Clinical Trials of UTD1 Injection Plus Capecitabine Versus Capecitabine Alone in Patients With Advanced and Metastatic Breast Cancer
Brief Title: Clinical Study of UTD1 Injection in Combination With Capecitabine in Patients With Advanced and Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Biostar Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BG01-1323L
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UTD1 Injection plus capecitabine (Experimental): UTD1 Injection: 30 mg/m2/day, IV on day 1-day 5 of each 21 day cycle; Capecitabine: 2000 mg/m2/day, oral bid on day 1-day 14 of each 21 day cycle.
  Number of Cycles: until progression or unacceptable toxicity develops.
  Interventions: Drug: UTD1 Injection plus capecitabine
- capecitabine (Active Comparator): Capecitabine: 2500 mg/m2/day, oral bid on day 1-day 14 of each 21 day cycle.
  Number of Cycles: until progression or unacceptable toxicity develops.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: UTD1 Injection plus capecitabine
  Arms: UTD1 Injection plus capecitabine
Drug: Capecitabine
  Arms: capecitabine

SUMMARY:
The purpose of this study is to determine whether UTD1 Injection in combination with capecitabine is effective in the treatment of advanced metastatic breast cancer using capecitabine as a control.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or cytologically diagnosed patients with advanced, metastatic breast cancer,or lacking standard therapy or being failed to or recurrent after standard therapy;
2. Patients who have previously treated with ≤4 chemotherapeutic regimes;
3. Patients who have previously treated with an anthracyclin antibiotics and a taxane;
4. Age 18 -70 years old, ECOG performance status of 0-2; Life expectancy of 3 months or more;
5. Patients with at least 1 measurable target lesion determined by CT within 2 weeks prior to enrollment;
6. Neuropathy <CTC2 degree （NCI CTC4.03）within 4 weeks prior to enrollment;
7. Basically normal results from routine blood test within 1 week prior to enrollment;
8. Basically normal liver and renal functions within 1 week prior to enrollment;
9. No abnormal function for major internal organs, no heart diseases.

Exclusion Criteria:

1. Received chemotherapy, radiotherapy, therapies with hormones or molecularly targeted drugs 4 weeks prior to enrollment, or received other chemotherapies while participating in this trial;
2. Patients with documented hypersensitivity to Cremophor EL, or patients with previous taxane treatment related SAE;
3. Patients of pregnancy or breast feeding;
4. Patients with previous standard capecitabine treatment ineffective, or patients received standard capecitabine treatment effective, but with less than 6 months of capecitabine clearance period;
5. Patients with uncontrolled brain metastasis or bone metastasis, which plan for recent surgery or local radiotherapy, or other emergency treatment;
6. Patients combined with severe and /or uncontrolled medical conditions, including severe cardiovascular disease, uncontrolled diabetes and high blood pressure, severe infection, severe gastrointestinal ulceration, and patients with incontrollable psychiatric history;
7. Patients with poor compliance;
8. Patients not fitted for this study determined by the investigators.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Progresssion free survival (PFS) | 2.0 years

SECONDARY OUTCOMES:
Overall survival (OS) | 4 years
Objective Response Rate(ORR） | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: B Xu, doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (11):
- China (11):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The Hospital Affiliated To Military Medical Science, Beijing, Beijing Municipality
  - The General Hospital of the People's Liberation Army, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - the First Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Xu B, Sun T, Zhang Q, Zhang P, Yuan Z, Jiang Z, Wang X, Cui S, Teng Y, Hu XC, Yang J, Pan H, Tong Z, Li H, Yao Q, Wang Y, Yin Y, Sun P, Zheng H, Cheng J, Lu J, Zhang B, Geng C, Liu J, Shen K, Yu S, Li H, Tang L, Qiu R; study group of BG01-1323L. Efficacy of utidelone plus capecitabine versus capecitabine for heavily pretreated, anthracycline- and taxane-refractory metastatic breast cancer: final analysis of overall survival in a phase III randomised controlled trial. Ann Oncol. 2021 Feb;32(2):218-228. doi: 10.1016/j.annonc.2020.10.600. Epub 2020 Nov 11. PMID 33188874
- [Derived] Xu J, Wang Y, Jiang C, Cao H, Jiang J, Xu B, Sun T. Ganglioside Monosialic Acid Alleviates Peripheral Neuropathy Induced by Utidelone Plus Capecitabine in Metastatic Breast Cancer From a Phase III Clinical Trial. Front Oncol. 2020 Oct 9;10:524223. doi: 10.3389/fonc.2020.524223. eCollection 2020. PMID 33163394
- [Derived] Zhang P, Sun T, Zhang Q, Yuan Z, Jiang Z, Wang XJ, Cui S, Teng Y, Hu XC, Yang J, Pan H, Tong Z, Li H, Yao Q, Wang Y, Yin Y, Sun P, Zheng H, Cheng J, Lu J, Zhang B, Geng C, Liu J, Peng R, Yan M, Zhang S, Huang J, Tang L, Qiu R, Xu B; BG01-1323L study group. Utidelone plus capecitabine versus capecitabine alone for heavily pretreated metastatic breast cancer refractory to anthracyclines and taxanes: a multicentre, open-label, superiority, phase 3, randomised controlled trial. Lancet Oncol. 2017 Mar;18(3):371-383. doi: 10.1016/S1470-2045(17)30088-8. Epub 2017 Feb 11. PMID 28209298